CLINICAL TRIAL: NCT01722214
Title: Randomized Multicenter Placebo-controlled Trial on the Effect of Adalumumab on Vascular Inflammation in Patient With Moderate to Severe Psoriasis
Brief Title: Trial on the Effect of Adalimumab on Vascular Inflammation in Patients With Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Abbott (Industry); Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Inno-6025
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Psoriasis; Vascular Inflammation; Coronary Atherosclerosis
Keywords: Psoriasis; Vascular Inflammation; Coronary Atherosclerosis; Ascending aorta; Pet scan; MRI
MeSH Terms: conditions — Psoriasis; Coronary Artery Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Adalimumab (Experimental): A total of 53 patients with moderate to severe psoriasis will randomized in the adalimumab group. At Day 0 patients will receive adalimumab. It will be administered sub-cutaneously as described in the Canadian product monograph (80mg followed by 40mg at Week 1 and 40mg every other week). At Week 16, all patients will received two injections of placebo. As of Week 17, patients randomized to the adalimumab group will receive 40 mg adalimumab every other week until Week 51.
  Interventions: Biological: Adalimumab
- Placebo Group (Placebo Comparator): A total of 53 patients with moderate to severe psoriasis will be randomized in the placebo group. At Day 0 these patients will receive the placebo. It will be administered sub-cutaneously as described in the Canadian product monograph of adalimumab. At Week 16, all these patients will received two injections of adalimumab. As of Week 17, patients randomized to the placebo group will receive 40 mg adalimumab every other week until Week 67.
  Interventions: Biological: Adalimumab; Other: Placebo

INTERVENTIONS:
Biological: Adalimumab — Injection of adalimumab (80 mg followed by 40 mg at week 1 and 40 mg EOW thereafter for 52 weeks). For Adalimibab group and Placebo group.
  Other Names: Humira
Other: Placebo — Injection of placebo that is physicaly identical to adalimumab without the active ingredient at identical intervals.
  Arms: Placebo Group

SUMMARY:
This study is a double-blinded randomized multicenter placebo controlled trial to determine the effect of adalimumab on vascular inflammation (ascending aorta and carotides) in patients with moderate to severe psoriasis.

DETAILED DESCRIPTION:
Patients with moderate to severe psoriasis will be included in this multicenter, double-blind, placebo controlled study. Patients will be randomized (1:1) at Day 0 to receive either adalimumab or placebo. Adalimumab will be administered sub-cutaneously as described in the Canadian product monograph (80mg followed by 40mg at Week 1 and 40mg every other week). At Week 16, all patients will receive two injections of blinded study products. Patients randomized to the placebo group will receive two injections of adalimumab (2 x 40 mg) and patients randomized to adalimumab will receive two injections of placebo. As of Week 17, patients randomized to the placebo group will receive 40 mg adalimumab every other week until Week 67. Patients randomized to the adalimumab group will continue to receive adalimumab 40mg every other week until Week 51.

Efficacy will be assessed with 18-FluoroDeoxyGlucose Positron Emission Tomography (FDG-PET) scan and carotid MRI at baseline, Week 16 and Week 52 (or Week 68 for patients randomized to placebo).

Safety will be assessed with physical examinations, vital signs, adverse events collection, routine laboratory examinations, pregnancy test, hepatitis B and C serology (screening), Purified Protein Derivative (PPD) or Quantiferon Gold (screening) and Chest X-Ray (CXR) (screening).

ELIGIBILITY:
Inclusion Criteria:

Patient has plaque psoriasis. Patient has at least a 6 month history of plaque psoriasis.Patient has a Body Surface Area (BSA) covered with psoriasis of 5% or more at Day 0.

Patient is a candidate for systemic therapy. Patient is male or female, 18 to 80 years of age at time of consent. Patient's weight at screening is a maximum of 180 kg. Patient using medication to control angina, hypertension, serum lipids and any medication that can have an effect on inflammation must be on a stable dose for at least 8 weeks before Day 0.

Patient has an ascending aorta atherosclerotic plaque inflammation target-to-background ratio of 1.6 or more as determined by 18-FDG uptake measured by PET scanning.

Patient or patient's partner has been in a menopausal state for at least a year, is surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation or vasectomy), is clinically diagnosed infertile, has a same-sex partner, is abstinent, or is willing to use effective contraceptive method for at least 30 days before Day 0 and at least 6 months after the last study drug administration. Effective contraceptive methods are:

1. Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream;
2. Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring;
3. Intrauterine device (IUD); Female patients of childbearing potential must have a negative serum pregnancy test at the Screening visit.

Patient is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination, and CXR performed at Screening.

Patient will be evaluated for latent TB infection with a PPD or a Quantiferon Gold test and CXR. Patient who demonstrates evidence of latent TB infection (either PPD more than or equal to 5 mm of induration or positive Quantiferon Gold, irrespective of Bacillus Calmette-Guerin (BCG) vaccination status and negative CXR findings for active TB, and/or suspicious CXR findings) will not be allowed to participate in the study.

Patient must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

Patient must be able and willing to self-administer SC injections or have a qualified person available to administer SC injections.

Exclusion Criteria:

Patient has spontaneously improving or rapidly deteriorating plaque psoriasis. Patient has other active infections (bacterial, fungal or viral) or skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis or with patient's safety.

Patient has a history of an allergic reaction or significant sensitivity to constituents of study drug, including latex (a component of the pre-filled syringe).

Patient has used a non-biological systemic therapy for the treatment of psoriasis less than 30 days before Day 0.

Patient has used an investigational chemical or biological agent less than 30 days or 5 half-lives prior to the Day 0 visit (whichever is longer).

Patient has used a biological therapy for the treatment of psoriasis less than 90 days before day 0.

Patient has used a systemic immnosuppressor (eg. Azathioprine, 6-mercaptopurine) less than 30 days before Day 0.

Patient is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.

Patient has used a topical treatment for psoriasis or has used phototherapy within the last 2 weeks prior to Day 0 (at the exception of low potency topical corticosteroids for groin, genitals, face, inflammatory area, palms and soles).

Patient has received Anakinra/Kineret within the last 2 weeks prior to the Day 0 visit or is likely to receive Anakinra/Kineret during the course of the study Patient has a poorly controlled medical condition, such as uncontrolled diabetes, documented history of recurrent infections, unstable ischemic heart disease, class III or IV (New York Heart Association Functional Classification; NYHA) congestive heart failure, an ejection fraction of less than 30%, recent stroke (within the past 3 months), chronic leg ulcer or any other condition which, in the opinion of the investigator, would put the patient at risk if participating in the study.

Patient has had a myocardial infarction or has been hospitalized for a cardiac condition within the past 12 weeks.

Patient has a history of acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft, carotid endarterectomy, stent installation or carotid revascularization within 12 weeks of Day 0.

Patient has had a percutaneous coronary intervention in the past 12 months. Patient plans for a change in medical treatment for angina, serum lipids, hypertension or any other medication that can have a significant effect on inflammation during the course of the study.

Patient has history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease (e.g. optic neuritis, visual disturbance, gait disorder/ataxia, facial paresis, apraxia).

Patient has history of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.

Patient has a history of listeriosis, treated or untreated Tuberculosis (TB), persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infectives within 30 days prior to the Day 0 visit or oral anti-infectives within 14 days prior to the Day 0 visit.

Patient has received a live attenuated vaccine 28 days or less before Day 0 or plan to receive a live attenuated vaccine during the study and up to 4 months after the last study drug administration..

Patient with hepatitis B or hepatitis C viral infection Patient with any of the following: hemoglobin ≤ 10 g/L, white blood cell count ≤ 3.0 X 109/L, platelet count ≤130 X 109/L, ALT ≥ 2 times the upper limit of normal, AST ≥ 3 times the upper normal limit, total bilirubin ≥ 2 times the upper normal limit or creatinine ≥ 150 µmol/L.

Patient currently uses or plans to use anti-retroviral therapy at any time during the study.

Patient is known to have immune deficiency or is immunocompromised. Female patient who is pregnant or breast-feeding or considering becoming pregnant during the study or for 6 months after the last dose of study medication.

Patient has a history of clinically significant drug or alcohol abuse in the last year.

Patient who plans to travel in an area where tuberculosis is endemic during the study and up to 4 months after the last study drug administration.

Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the target (atherosclerotic plaque) to background (blood) ratio (TBR) from the ascending aorta at Week 16 for patients randomized to adalimumab as compared to patients randomized to placebo | Baseline, Week 16 and Week 52 or 68

SECONDARY OUTCOMES:
Change from baseline in the TBR from the mean of both carotid arteries at Week 16 for patients randomized to adalimumab as compared to patients randomized to placebo | Baseline, Week 16 and Week 52 or 68
Change from baseline in the TBR from the ascending aorta 52 weeks after the first dose of adalimumab | Baseline and Week 52 or 68
Change from baseline in the TBR from the mean of both carotid arteries 52 weeks after the first dose of adalimumab | Baseline and Week 52 or 68
Change from baseline in carotid wall area at Week 16 as measured by MRI for patients randomized to adalimumab as compared to patients randomized to placebo | Baseline and Week 16
Change from baseline in carotid wall area as measured by Magnetic Resonance Imaging (MRI) 52 weeks after the first dose of adalimumab | Baseline and Week 52 or 68
Change from baseline in hsCRP at Week 16 for patients randomized to adalimumab as compared to patients randomized to placebo | Baseline and Week 16
Change from baseline in serum lipids (total cholesterol, LDL- calc, HDL cholesterol, triglycerides) at Week 16 for patients randomized to adalimumab as compared to patients randomized to placebo | Baseline, Week 16
Correlation between change from baseline in TBR from the ascending aorta at Week 16 and change from baseline in PASI at Week 16 | Baseline and Week 16
Correlation between change from baseline in PASI at Week 16 and change in hsCRP at Week 16 | Baseline and week 16
Correlation between change from baseline in TBR from the ascending aorta at Week 16 and change from baseline in hsCRP at Week 16 | Baseline and Week 16
Correlation between change from baseline in TBR at Week 16 from the ascending aorta and change from baseline in skin inflammation as measured by PET-Scan at Week 16 | Baseline and Week 16

OTHER OUTCOMES:
Change from baseline in hsCRP protein levels at 52 weeks after the first dose of adalimumab | Baseline and Week 52 or 68
Change from baseline in serum lipids (total cholesterol, LDL- calc, HDL cholesterol, triglycerides) 52 weeks after the first dose of adalimumab | Baseline and Week 52 or 68

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research; Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (5):
- Canada (5):
  - Lynderm Research Inc., Markham, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Montreal Healt Institute, Montreal, Quebec
  - Innovaderm Research Inc, Montreal, Quebec
  - Clinique Médicale Dr Isabelle Delorme, Saint-Hyacinthe, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelfand JM, Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB. Risk of myocardial infarction in patients with psoriasis. JAMA. 2006 Oct 11;296(14):1735-41. doi: 10.1001/jama.296.14.1735. PMID 17032986
- [Background] Gelfand JM, Dommasch ED, Shin DB, Azfar RS, Kurd SK, Wang X, Troxel AB. The risk of stroke in patients with psoriasis. J Invest Dermatol. 2009 Oct;129(10):2411-8. doi: 10.1038/jid.2009.112. Epub 2009 May 21. PMID 19458634
- [Background] Prodanovich S, Kirsner RS, Kravetz JD, Ma F, Martinez L, Federman DG. Association of psoriasis with coronary artery, cerebrovascular, and peripheral vascular diseases and mortality. Arch Dermatol. 2009 Jun;145(6):700-3. doi: 10.1001/archdermatol.2009.94. PMID 19528427
- [Background] Miyasaka Y, Barnes ME, Petersen RC, Cha SS, Bailey KR, Gersh BJ, Casaclang-Verzosa G, Abhayaratna WP, Seward JB, Iwasaka T, Tsang TS. Risk of dementia in stroke-free patients diagnosed with atrial fibrillation: data from a community-based cohort. Eur Heart J. 2007 Aug;28(16):1962-7. doi: 10.1093/eurheartj/ehm012. Epub 2007 Apr 25. PMID 17459900
- [Background] van Leuven SI, Franssen R, Kastelein JJ, Levi M, Stroes ES, Tak PP. Systemic inflammation as a risk factor for atherothrombosis. Rheumatology (Oxford). 2008 Jan;47(1):3-7. doi: 10.1093/rheumatology/kem202. Epub 2007 Aug 16. PMID 17702769
- [Background] Mehta NN, Yu Y, Saboury B, Foroughi N, Krishnamoorthy P, Raper A, Baer A, Antigua J, Van Voorhees AS, Torigian DA, Alavi A, Gelfand JM. Systemic and vascular inflammation in patients with moderate to severe psoriasis as measured by [18F]-fluorodeoxyglucose positron emission tomography-computed tomography (FDG-PET/CT): a pilot study. Arch Dermatol. 2011 Sep;147(9):1031-9. doi: 10.1001/archdermatol.2011.119. Epub 2011 May 16. PMID 21576552
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Moubayed SP, Heinonen TM, Tardif JC. Anti-inflammatory drugs and atherosclerosis. Curr Opin Lipidol. 2007 Dec;18(6):638-44. doi: 10.1097/MOL.0b013e3282f0ee11. PMID 17993809
- [Background] Dixon WG, Symmons DP. What effects might anti-TNFalpha treatment be expected to have on cardiovascular morbidity and mortality in rheumatoid arthritis? A review of the role of TNFalpha in cardiovascular pathophysiology. Ann Rheum Dis. 2007 Sep;66(9):1132-6. doi: 10.1136/ard.2006.063867. Epub 2007 Jan 24. PMID 17251223
- [Background] Jacobsson LT, Turesson C, Gulfe A, Kapetanovic MC, Petersson IF, Saxne T, Geborek P. Treatment with tumor necrosis factor blockers is associated with a lower incidence of first cardiovascular events in patients with rheumatoid arthritis. J Rheumatol. 2005 Jul;32(7):1213-8. PMID 15996054
- [Background] Dixon WG, Watson KD, Lunt M, Hyrich KL; British Society for Rheumatology Biologics Register Control Centre Consortium; Silman AJ, Symmons DP; British Society for Rheumatology Biologics Register. Reduction in the incidence of myocardial infarction in patients with rheumatoid arthritis who respond to anti-tumor necrosis factor alpha therapy: results from the British Society for Rheumatology Biologics Register. Arthritis Rheum. 2007 Sep;56(9):2905-12. doi: 10.1002/art.22809. PMID 17763428
- [Background] Turesson C, McClelland RL, Christianson TJ, Matteson EL. Severe extra-articular disease manifestations are associated with an increased risk of first ever cardiovascular events in patients with rheumatoid arthritis. Ann Rheum Dis. 2007 Jan;66(1):70-5. doi: 10.1136/ard.2006.052506. Epub 2006 Jul 28. PMID 16877533
- [Background] Wu F. The effect of tumor necrosis factor-alfa inhibitors on the risk of myocardial infarction in patients with psoriasis. E-poster session presented at the 69th American Academy of Dermatology, Abstract P400; 4-8 Feb 2011; New Orleans, USA.
- [Background] Davidovici BB, Sattar N, Prinz J, Puig L, Emery P, Barker JN, van de Kerkhof P, Stahle M, Nestle FO, Girolomoni G, Krueger JG. Psoriasis and systemic inflammatory diseases: potential mechanistic links between skin disease and co-morbid conditions. J Invest Dermatol. 2010 Jul;130(7):1785-96. doi: 10.1038/jid.2010.103. Epub 2010 May 6. PMID 20445552
- [Background] Ko H-S, M.D. Medical Officer, Division of Dermatologic and Dental Drug Products, Center for Drug Evaluation and Research, Food and Drug Administration, Bethesda MD. Clinical Design for Psoriasis [presentation]. Dermatologic and Ophthalmic Drugs Advisory Committee 49th Meeting Open Session (Volume II); Gaithersburg, MD. 1998 March 20.
- [Background] Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44. doi: 10.1159/000250839. PMID 357213
- [Background] Marks R, Barton SP, Shuttleworth D, Finlay AY. Assessment of disease progress in psoriasis. Arch Dermatol. 1989 Feb;125(2):235-40. PMID 2643928
- [Background] Ahlehoff O, Gislason GH, Lindhardsen J, Olesen JB, Charlot M, Skov L, Torp-Pedersen C, Hansen PR. Prognosis following first-time myocardial infarction in patients with psoriasis: a Danish nationwide cohort study. J Intern Med. 2011 Sep;270(3):237-44. doi: 10.1111/j.1365-2796.2011.02368.x. Epub 2011 Mar 24. PMID 21362070
- [Derived] Bissonnette R, Harel F, Krueger JG, Guertin MC, Chabot-Blanchet M, Gonzalez J, Maari C, Delorme I, Lynde CW, Tardif JC. TNF-alpha Antagonist and Vascular Inflammation in Patients with Psoriasis Vulgaris: A Randomized Placebo-Controlled Study. J Invest Dermatol. 2017 Aug;137(8):1638-1645. doi: 10.1016/j.jid.2017.02.977. Epub 2017 Mar 9. PMID 28286061